CLINICAL TRIAL: NCT05182086
Title: IMPROVE: Evaluation of a Combined Lifestyle Intervention Program to Improve Quality of Life in Long-term ICU-survivors
Brief Title: Improving Recovery After Critical Illness
Acronym: IMPROVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University of Groningen (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Principle Investigator, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTPO 1103
Record Dates: First submitted 2021-08-31; First posted 2022-01-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Post Intensive Care Unit Syndrome; Critical Illness; Malnutrition; Muscle Weakness
MeSH Terms: conditions — Critical Illness; Malnutrition; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients that are allocated to the intervention group will participate in a 12 week lifestyle intervention program consisting of group exercise therapy and dietary advice combined with dietary supplementation. The group exercise therapy will be guided by trained physical therapists. Patients will participate in this part of the intervention twice a week for one hour. The exercise therapy will combine cardiorespiratory with strength training. At the start of the intervention, patients will have an appointment with a nutritional scientist or doctor in which they will receive dietary advise and dietary supplements (ProSource®) to reach the advised caloric and protein intake as composed by the Dutch Centre for Nutrition (Voedingscentrum). Dietary supplements like ProSource® are extensively tested and often used as part of general practice to patients after ICU- or hospital-discharge following critical illness.
  Interventions: Other: Group physical therapy and dietary improvements
- Standard care (No Intervention): Standard care outpatient post-ICU clinic

INTERVENTIONS:
Other: Group physical therapy and dietary improvements — 20 patients allocated to intervention group. During 12 weeks, patients will participate in a combined lifestyle intervention, including a one-hour physical therapist guided exercise group twice a week and consultation by a nutritional scientist. In case of inadequate intake, dietary supplements will be provided.
  Arms: Intervention group

SUMMARY:
Rationale: Survival rates of patients with critical illness have increased due to improved facilities and treatment methods in the intensive care unit (ICU). However, surviving critical illness does not mean these patients are cured. In general, ICU-admission is associated with decreased physical performance and perceived physical health, impaired mental health and quality of life (QoL), reflecting in an impaired long-term recovery. Long-term health problems can partly be contributed to prolonged muscle weakness and malnutrition. Improving physical performance and perceived physical health may play a key role in boosting recovery after ICU-admission. Mono-interventions focusing on improving physical performance or nutritional intake have limited effect on long term functioning and QoL. A lifestyle intervention encompassing physical therapy and optimisation of caloric and protein intake may improve wellbeing and QoL in these patients. Previous studies found that interventions focused on mobilization and physical rehabilitation are feasible within the ICU and outpatient programs. Additionally, promising results were found in personalized healthcare and lifestyle programs for other patient groups with long-term health problems, such as cancer survivors and patients with diabetes or mental health problems. Based on this, the investigators hypothesized that a lifestyle intervention program may improve wellbeing and quality of life in long-term ICU-survivors.

Objective: Evaluation of the effects of a integrative lifestyle intervention program on physical performance and perceived physical health, mental health and health related quality of life after ICU-admission.

Study design: Randomised controlled trial Study population: Long-term ICU patients (length of stay ICU ≥48h) Intervention: The intervention group will be part of a 12-week combined lifestyle intervention encompassing group physical therapy twice a week and improvement of dietary caloric and protein intake by means of nutritional advice and, if applicable, caloric and/or protein supplementation. The control group will be subject to follow up meetings with research staff to assess physical and mental health and quality of life.

Main study parameters/endpoints: Physical functioning (RAND-36 subscale-score) at the end of the 12 week intervention period.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants have two additional appointments where they participate in an interview and perform physical tests (bioimpedance measurements, ultrasound of the upper thigh muscles, hand grip strength test, Morton mobility index test, and the six-minute walking test with pulse oximetry). At baseline and week 12 of the program, all participants complete a combination of questionnaires on mental health and quality of life. The intervention group will additionally be subject to supervised group training sessions twice a week for the duration of the intervention (12 weeks). Further, two meetings with a professional about their diet will be organised. If a patient has a deficit in caloric and/or protein intake, dietary supplements with daily intake instructions will be provided. The risks and disadvantages of this intervention are minimal. However, this study requires considerable time investment and physical and mental effort. The extent of this study is crucial to clarify the effect of a combined intervention program on recovery after critical illness.

DETAILED DESCRIPTION:
Survival rates of critical illness have increased due to improved facilities and treatment methods in intensive care units. However, surviving critical illness does not automatically mean these patients are cured. In the past, the patients' survival was the measure of success in the treatment of critical illness. Over the past decades, the focus has been shifting towards the quality of life and care needs of these patients after critical illness. Survivors of critical illness frequently suffer from reduced quality of life. Health problems in the recovery period of survivors may predominantly be provoked by the physical consequences of longterm ICU-admission. The physical consequences of critical illness are mostly associated with skeletal muscle wasting during critical illness. This results in a decrease of muscle density up to two percent per day. Some long term physical health problems associated with this phenomenon are fatigue, neuropathy, neuromuscular dysfunction, and changes in bone mineral density. With regards to the long term psychosocial problems in survivors of critical illness there have been reports of short and long-term anxiety, depression and/or posttraumatic stress disorder (PTSD). Further, during and after critical illness, patients may experience delirium and cognitive impairments. In conclusion, survivors of critical illness suffer from long term physical and mental health problems, reflecting in a reduced HRQoL.

Critical illness survivorship is a relatively new and unknown area in research and medical health care. The term post-intensive care syndrome (PICS) has been used to describe the complex aetiology of health deficits following critical illness. A recent Dutch study (the MONITOR-IC-study) with a population of 1729 ICU-patients found that an overwhelming 70 percent of ICU-patients suffer from some form of PICS one year after discharge. Data collected from the specialized post-ICU clinic of the Medical Centre Leeuwarden (MCL) illustrated that 44% of 250 patients that visited this clinic between 2012 and 2018 were unable to sufficiently recover in physical functioning one year after ICU-discharge. Unfortunately, adequate and efficient aftercare programs for ICU survivors are still lacking and patients regularly feel abandoned and insecure after discharge. Personalised healthcare and lifestyle interventions may fulfil this discontinuity in care and improve physical performance and perceived physical health in ICU-patients, followed by improvements in mental wellbeing and HRQoL. Little is known on the effects of optimizing lifestyle on longterm recovery of these patients. Promising results were found in personalised healthcare and lifestyle programs for other patient groups with long-term health problems, such as cancer survivors and patients with diabetes or mental health problems. A Cochrane review showed several exercise rehabilitation programs after ICU-discharge to be feasible, but lacking in overall effect on functional exercise capacity, or on health-related quality of life. This paucity of effect on patient-centred outcomes may be due to inconsistencies in study protocol. However, a lack of adequate nutritional support might be an equally important pitfall. ICU-survivors may experience a number of problems that can hinder their nutritional intake, including lack of appetite, problems with taste and smell perception, and swallowing issues. Recent data from a study on post-ICU nutritional intake showed that of 12 included patients, the majority did not meet their daily caloric and protein intake. Data on nutritional intake after hospital discharge is lacking, but it is likely that patients are unable to achieve these goals without professional support.

Based on this, the investigators hypothesized that, complementary to the standard post-ICU care, a combined lifestyle intervention focussed on exercise and nutritional therapy may improve physical performance and perceived physical health alongside with an improved mental wellbeing and quality of life in long-term ICU-survivors.

ELIGIBILITY:
Inclusion criteria Long stay post-ICU patients (length of stay ≥48h) between 6 weeks and 6 months after hospital discharge AND >18 years old AND able to visit the hospital 2 times a week AND a RAND-36 physical functioning subscale score < 67%

Exclusion criteria

* Allergy to components of ProSource® (Allergy information: gluten-free, lactose-free, NOT cow's milk free (wey-protein), produced in a factory in which soy, wheat and nuts are processed.
* Inability to understand the Dutch language
* Actively participating in a professional physical rehabilitation program during the study period.

Note: previous participation in a concluded rehabilitation program is NOT an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | After the 12-week intervention program
  Physical functioning (subscale score) measured with the Dutch 36-Item Short Form health Survey/Research and Development-36 (RAND-36) questionnaire (0-100; higher is better)

SECONDARY OUTCOMES:
Change in hand grip strength | Before and after the 12-week intervention program
  Hand grip strength with hand-held dynamometer (kg; higher is better)
Change in walking distance | Before and after the 12-week intervention program
  Walking distance with the six-minute walking test (m, higher is better)
Change in quadriceps muscle layer thickness | Before and after the 12-week intervention program
  Ultrasound measures of the quadriceps (mm, higher is better)
Change in mobility | Before and after the 12-week intervention program
  Mobility using the morton mobility index (0-100, higher is better)
Change in dietary intake | Before and after the 12-week intervention program
  Dietary intake using food diary
Change in health-related quality of life | Before and after the 12-week intervention program
  Dutch 36-Item Short Form health Survey/Research and Development-36 (RAND-36) questionnaire (0-100; higher is better)
Change in fatigue | Before and after the 12-week intervention program
  Short Fatigue Questionnaire (Verkorte VermoeidheidsVragenlijst) (4-28, higher is worse)
Change in anxiety and depression symptoms | Before and after the 12-week intervention program
  Hospital Anxiety and Depression Scale (HADS) (0-21; higher is worse)
Change in cognitive functioning | Before and after the 12-week intervention program
  Cognitive Failure Questionnaire (CFQ) (0-100; higher is worse)
Change in subjective happiness | Before and after the 12-week intervention program
  Happiness Index (HI) VAS-scale (0-10; higher is better)
Phase angle | Before and after the 12-week intervention program
  Bioimpedence measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided